CLINICAL TRIAL: NCT02643069
Title: Feasibility and Effectiveness of Frailty Screening and Management Programs Implemented in Different Clinical Settings (FRAILCLINIC)
Brief Title: Clinical Intervention in Frail Older People (FRAILCLINIC)
Acronym: FRAILCLINIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20131208
Record Dates: First submitted 2015-03-26; First posted 2015-12-30 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Frailty Syndrome
Keywords: Frailty; Frailty tools; Clinical settings; Disability; Quality of life; Functional Autonomy
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Geriatric Program (Experimental): A comprehensive management plan of the frail patients, covering both in-hospital and postdischarge time, according to the treating physicians (s) surgeon and the performance of a geriatrician . This management will consist of the therapeutic plan, access to geriatric levels of care, coordination with primary and social care, rehabilitation, and discharge plan.
  Interventions: Other: Intervention Geriatric Program
- Usual clinical practice (No Intervention): A comprehensive management plan of the frail patients, covering both in-hospital and postdischarge time, agreed with the treating physicians (s) surgeon.

INTERVENTIONS:
Other: Intervention Geriatric Program — The investigators will implemented programs to detected and manage care for older patients in four settings: Emergency room, oncology department, surgery departments making major surgery and Cardiology. The core intervention will consist of the following elements: comprehensive geriatric assessment, coordination with primary ans social care, integrated and continued care, access to rehabilitation facilities, management of drug treatment avoiding polypharmacy and stressing adherence.
  Arms: Intervention Geriatric Program

SUMMARY:
Frailty is the main risk factor for the development of incident disability in older people and one of the most important for other adverse outcomes (death, hospitalisation, falls, and permanent institutionalisation).

Although frailty is a frequent condition in older adults who attend hospitals, little is known about its true prevalence in different settings of care. Better knowledge of this issue will inform the rational design of more effective strategies aimed at providing fitted care for these patients. Thus, the current study will potentially have impact on the quality of care for frail patients by revealing the prevalence of frailty in different settings of care, the difficulties in detection and management of frailty in these settings and the best instruments to detect frailty.

The investigators proposal brings together 6 partners in the European Union (EU) from three countries, with the common aim of studying the feasibility of a program to detect frail older patients in high risk clinical settings.

DETAILED DESCRIPTION:
Quality assurance plan:

* To perform regular monitoring according to the International Conference on Harmonisation (ICH) and Good Clinical Practice (GCP): The data will be evaluated according to the protocol and source documents.
* To give training to the centres involved in the study.
* To check the electronic Case Report Form (eCRF)

Data checks to compare data entered into the registry:

The eCRF has been designed to capture all data required in the protocol. A unique eCRF will be completed for subject, taking into account the protection law in each country of the study.Subjects will be identified by a unique subject number (with key held by the relevant partner), so none id card number will not be recorded on the eCRF or the database. The monitor will guarantee that the eCRF is fully and correctly fill up according to the source documents. The researcher will assure that all data recorded in the eCRF coincide with the information recorded in the source documents.

Plan for missing data to address situations where variables are reported as missing:

The investigators will check the missing data in each eCRF and source documents.

Statistical analysis:

Data will be analyzed using STATA®. Descriptive statistics will be reported and histograms will assess the distribution of frailty scores in each scale. Each analysis will be categorised according to frail, prefrail or robust patients.The prevalence of frailty will be calculated for each scale based on the score thresholds and relationships between frailty and age and other variables will be evaluated. Agreement among scales will be examined using the Cohen kappa statistic. Receiver operator characteristic (ROC) curves will be constructed to compare the area under the ROC curve (AUC) for each scale for available outcomes.

Sample Size: A minimum of 50 patients will be studied in each clinical setting, providing a database of 900 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Frailty patients older than 75 years old attended in the settings of care.
2. Willing and able to provide informed consent

Exclusion Criteria:

1. Lack of capacity to give informed consent.
2. Those unable or unwilling to cooperate with any of the assessments

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 821 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Functional Status assessed using the Barthel index for Basic Activities of Daily Living | 36 months
  will be assessed using the Barthel index for Basic Activities of Daily Living
Functional Status assessed using the Lawton index for Instrumental Activities of Daily Living | 36 months
  will be assessed using the Lawton index for Instrumental Activities of Daily Living
Institutionalization (defined as the number of patients newly addressed to nursing) | 36 months
  defined as the number of patients newly addressed to nursing
Mortality | 36 months
  number of deaths occurred either during hospitalization or at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Leocadio Rodriguez Mañas, IP, Principal Investigator — Hospital Universitario de Getafe
Locations (1):
- Hopsital Universitario de Getafe, Getafe, Madrid, Spain

REFERENCES:
- [Background] Rodriguez-Manas L, Fried LP. Frailty in the clinical scenario. Lancet. 2015 Feb 14;385(9968):e7-e9. doi: 10.1016/S0140-6736(14)61595-6. Epub 2014 Nov 6. No abstract available. PMID 25468154
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Result] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Result] Pena FG, Theou O, Wallace L, Brothers TD, Gill TM, Gahbauer EA, Kirkland S, Mitnitski A, Rockwood K. Comparison of alternate scoring of variables on the performance of the frailty index. BMC Geriatr. 2014 Feb 24;14:25. doi: 10.1186/1471-2318-14-25. PMID 24559204
- [Result] Drubbel I, Numans ME, Kranenburg G, Bleijenberg N, de Wit NJ, Schuurmans MJ. Screening for frailty in primary care: a systematic review of the psychometric properties of the frailty index in community-dwelling older people. BMC Geriatr. 2014 Mar 6;14:27. doi: 10.1186/1471-2318-14-27. PMID 24597624
- [Result] Theou O, Brothers TD, Mitnitski A, Rockwood K. Operationalization of frailty using eight commonly used scales and comparison of their ability to predict all-cause mortality. J Am Geriatr Soc. 2013 Sep;61(9):1537-51. doi: 10.1111/jgs.12420. Epub 2013 Aug 26. PMID 24028357
- [Result] Morley JE, Malmstrom TK, Miller DK. A simple frailty questionnaire (FRAIL) predicts outcomes in middle aged African Americans. J Nutr Health Aging. 2012 Jul;16(7):601-8. doi: 10.1007/s12603-012-0084-2. PMID 22836700

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-08-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT02643069/Prot_SAP_ICF_000.pdf